CLINICAL TRIAL: NCT03558113
Title: Reliability of Secondary Caries Detection Around Composite Restoration Using Light Induced Fluorescence in Comparison to Visual Tactile Method: Diagnostic Accuracy Study
Brief Title: Reliability of Secondary Caries Detection Around Composite Restoration Using Light Induced Fluorescence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haneen ahmed shafik elmoselhy, master student, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEBD-CU-2018-06-04
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-06

CONDITIONS: Secondary Caries

STUDY DESIGN:
Intervention Model Description: Screening of patients that come to the conservative dentistry department seeking dental care will continue until the target population is achieved. The patients' restorations will be subjected to visual examination and diagnosis using dental charts. Once the patients that are potentially eligible for this study are identified, they will be contacted by the research investigator who will explain the study and ascertains the patient's interest. If interested, more detailed evaluations and preparations are made.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- visual tactile method (Other): visual tactile method using the modified USHPS critiria
  Interventions: Diagnostic Test: light induced fluorescence intraoral camera

INTERVENTIONS:
Diagnostic Test: light induced fluorescence intraoral camera — intraoral oral light induced fluorescence diagnostic camera
  Other Names: soprolife camera

SUMMARY:
A total of 29 volunteer patients will be assigned in this study. Each patient should have one resin composite restoration. The restoration will be evaluated by two diagnostic methods (D), where D1 represents visual-tactile assessment method (modified USPHS) and D2 represents light induced fluorescence intraoral camera

DETAILED DESCRIPTION:
Three operators, the researcher and the 2 supervisors, from the Conservative Dentistry Department, Faculty of Dentistry, Cairo University, will be the examiners in this study. Each examiner will record the dental findings using both the visual- tactile assessment method and the fluorescent-aided identification method. The visual-tactile assessment method includes the use of mirror, probe under good illumination condition, while the fluorescent-aided identification method will be performed by light induced fluorescence intraoral camera

ELIGIBILITY:
Inclusion Criteria:

* Patients should be over 18 years of age. Patients should have an acceptable oral hygiene level. Patients must have at least one posterior resin composite restoration

Exclusion Criteria:

Patients with a compromised medical history. Severe or active periodontal disease. Heavy bruxism or a traumatic occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
reliability and reproducibility of intra oral light fluorescence camera using kappa strength | 6 months
  in secondary craies diagnosis around composite restorations

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided